CLINICAL TRIAL: NCT02599675
Title: Effects of 12 Weeks of Vitamin D Supplementation on Muscle Characteristics in Trained Subjects
Brief Title: Vitamin D Supplementation and Muscle Characteristics in Trained Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Trainsome 2015#006
Record Dates: First submitted 2015-11-05; First posted 2015-11-06 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-03

CONDITIONS: Healthy Subjects, Trained
Keywords: Muscle; Vitamin D; Strength; Endurance; Muscle fiber
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Vitamin D3 capsules for 12 weeks (2000 IU daily, equivalent to 50 ug)
  Interventions: Dietary Supplement: Vitamin D3
- Placebo (Placebo Comparator): Placebo capsules for 12 weeks (the number of daily capsules will match that of the vitamin D-group)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 dissolved in olive oil, encapsuled
  Other Names: cholecalciferol
  Arms: Vitamin D3
Dietary Supplement: Placebo — Olive oil, encapsuled
  Arms: Placebo

SUMMARY:
This study evaluates the effect of vitamin D supplementation on outcomes muscle performance and characteristics in 70 trained healthy individuals (18-40 years of age). Subjects will be allocated to ingest either vitamin D (35) or placebo (35) in a double-blinded fashion

DETAILED DESCRIPTION:
Vitamin D insufficiency compromises muscle functionality, leading to changes in muscle mass and strength, manifested at the cellular level. While this is increasingly recognized as a problem for individuals with vitamin D deficiency (typically 25(OH)D < 25 nmol/l), there is no general consensus for the remainder of the vitamin D-spectra. This lack of knowledge is probably linked to the variation in protocols of studies that have investigated the physiological role of vitamin D. These variations vary from aspects such as interventional vs observational studies to aspects related to subject characteristics such as age, health and training status. In this project, we will evaluate the effects of 12 weeks of vitamin D supplementation (2000 IU/day) on muscle performance and characteristics in 70 trained healthy individuals (18-40 years of age). Subjects will be allocated to either a vitamin D (35) or a placebo group (35) in a double-blinded manner. They will be instructed to continue their ordinary modes and frequency of training.

We anticipate baseline vitamin D levels in blood (and hence changes in vitamin D obtained through supplementation), measured as 25(OH)D, to be a major determinant of the efficacy of the intervention. This means that we expect individuals with low baseline levels of 25(OH)D to display more pronounced changes in functional and biological outcome measures than those with high baseline values. Such a scenario could be related to an inability of our protocol to increase blood levels of 25(OH)D in individuals with higher physiological levels of vitamin D (which essentially means that ingestion of vitamin D3 is leveled out or exceeded by elimination of vitamin D derivatives). Alternatively, it may be related to inabilities of tissues to respond to the resulting elevation in vitamin D levels. To study the individual variation in vitamin D responses, data on both functional and biological variables will be divided into quartiles based on baseline 25(OH)D-levels, whereupon comparisons will be made between the low-end and high-end quartile. Individual variation will also be assessed using a mixed model approach.

ELIGIBILITY:
Inclusion Criteria:

- Individuals that have performed strength and / or endurance exercise training at least 3 X week for at least 6 months prior to the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-11; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Lower body maximal dynamic strength | wk 0, wk12
  Changes in the ability of lower body muscles to exert maximal force during a dynamic movement
Muscle fiber composition | wk0, wk12
  Changes of the muscle fiber composition of musculus vastus lateralis in a 2X to 2A direction, measured using mRNA profiling

SECONDARY OUTCOMES:
Gene expression in muscle | wk0, wk12
  Changes in RNA abundances in musculus vastus lateralis, measured at the level of single genes
Vitamin D in blood | wk0, wk12
  Changes in levels of 25(OH)D in blood
Steroid hormones in blood | wk0, wk12
  Changes in levels of steroid hormones in blood
Muscular endurance | wk0, wk12
  Changes in the ability of muscles to perform repeated dynamic contractions at submaximal loads (50% of 1 repetition maximum)
Upper body maximal dynamic strength | wk0, wk12
  Changes in the ability of upper body muscles to exert maximal force during dynamic movements

OTHER OUTCOMES:
Training diary | From 1 month prior to study to post test (w12)
  Diary that includes information on type of training, duration and intensity performed
Vitamin D-intake diary | From 1 month prior to study to post test (w12)
  Diary withthat includes information on approximate intake of vitamin D from sources other than the study-specific supplement, including ingestion of fish, seafood and vitamin D-supplement
Sun exposure diary | From 1 month prior to study to post test (w12)
  Diary that includes information on exposure to solarium or sun in countries south of Norway

CONTACTS AND LOCATIONS:
Overall Officials: Håvard Nygaard, MSc, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Lillehammer University College, Lillehammer, Norway